CLINICAL TRIAL: NCT04434612
Title: Effect of OXSIGHT Smart Glasses on Patients With Advanced Glaucoma
Acronym: OXSIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zhongshanOCOXSIGHT
Record Dates: First submitted 2020-06-10; First posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Advanced Glaucoma
Keywords: OXSIGHT; advanced glaucoma; low vision aids; head-mounted electronic devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OXSIGHT smart glasses (Experimental): Wearing OXSIGHT smart glasses
  Interventions: Device: OXSIGHT smart glasses

INTERVENTIONS:
Device: OXSIGHT smart glasses — OXSIGHT smart glasses are head-mounted electronic LVAs designed for LV patients with visual field loss.
  Other Names: There is no

SUMMARY:
Glaucoma is the leading cause of irreversible blindness worldwide. The visual function of patients with advanced glaucoma is severely impaired, and the vision-related activities (e.g. movement, reading) are obviously restricted, which may have a negative impact on the patients' quality of life (QOL) and increase the burden on individuals and families. Low vision aids (LVAs) and other devices for vision rehabilitation (VR) are useful for patients with advanced glaucoma to maximize the function of residual vision and improve the QOL. OXSIGHT smart glasses are the latest LVAs eyeglasses that are expected to improve the QOL for patients with low vision (LV), such as those with glaucoma. Clinical data were collected to evaluate the efficacy and its influencing factors of OXSIGHT smart glasses in patients with advanced glaucoma, in providing theoretical basis for subsequent clinical studies.

DETAILED DESCRIPTION:
1. Glaucomatous low vision. Glaucoma is a chronic eye disease that causes irreversible damage to the optic nerve and can lead to severe vision loss and blindness. Low vision (LV) is a decrease in vision that cannot be corrected with standard glasses, contact lenses, medication or surgery, impairing a person's ability to perform age-appropriate vision-dependent tasks.
2. Low vision rehabilitation. Low Vision Rehabilitation (LVR) is part of the continuum of eye care that extends from diagnosis to treatment and rehabilitation, designed to help visually impaired patients retain vision to the maximum, make activities easier to perform, regain independence, and improve their QOL. LVR services include comprehensive assessment of visual function, prescription of LVAs, rehabilitation training and referrals to a range of community services and psychosocial support.
3. Research status of intelligent head-mounted devices. In recent years, video head-mounted devices have been gradually applied in the field of VR, with the advantages of high definition, diverse processing modes, adjustable magnification, contrast and brightness, which overcome the limitations of traditional devices, like eSight 3, NuEyes, and IrisVision. However, studies on the effectiveness of head-mounted electronic LVAs are quite limited.
4. OXSIGHT smart glasses. OXSIGHT smart glasses, the latest generation of head-mounted electronic LVAs, developed by the team of Oxford University in the UK, are designed for LV patients with visual field defects. Based on the previous generation, OXSIGHT has the advantages of lighter weight, comfortable wearing, better imaging quality, multi-mode assisted visual recognition and so on. However, the efficacy and influencing factors of OXSIGHT smart glasses on advanced glaucoma patients remain unclear, and further studies are needed.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥10 years, able to complete all tests and inspections;
2. a definite diagnosis of primary or secondary glaucoma or glaucoma in children;
3. the best corrected visual acuity of the better eye is no more than 0.3 and better than 0.05; visual field ≤10° and MD value < -12db;
4. Visual acuity, intraocular pressure, and other eye conditions have been stable for more than 6 months.

Exclusion Criteria:

1. unable to cooperate with related inspections;
2. a history of eye surgery or eye laser within 6 months;
3. diseases that interfere with the diagnosis of glaucoma, such as optic disc dysplasia, obvious anisometropia, retinal vascular diseases, optic nerve diseases, macular degeneration, cerebrovascular diseases, etc.;
4. pregnant or lactating women;
5. those who refuse to sign the informed consent or voluntarily withdraw from the study due to discomfort or other reasons.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-06 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline CLVQOL scores at different time points | The examination was performed at 1 day, 1 week, 2 weeks, 4 weeks and 8 weeks after intervention.
  The Low vision Quality of Life Questionnaire (LVQOL) specifically investigates the QOL of visually impaired patients. The questionnaire consists of 25 closed items and examines four dimensions: distance vision, mobility and lighting; adjustment; reading and fine work; daily activities. As a convenient tool, LVQOL is widely used in clinical settings to evaluate effects of clinical treatment and corresponding strategies of low-vision rehabilitation. CLVQOL is the Chinese version of LVQOL.

SECONDARY OUTCOMES:
Changes from baseline visual acuity at different time points | The examination was performed at 1 day, 1 week, 2 weeks, 4 weeks and 8 weeks after intervention.
  ETDRS visual acuity chart was used.
Changes from baseline contrast sensitivity at different time points | The examination was performed at 1 day, 1 week, 2 weeks, 4 weeks and 8 weeks after intervention.
  Pelli-Robson Contrast Sensitivity Charts were used.
Changes from baseline visual field at different time points | The examination was performed at 1 day, 1 week, 2 weeks, 4 weeks and 8 weeks after intervention.
  Visual field was measured by the kinetic perimetry test of Humphrey field analyzer.
Changes from baseline scores of mobility test at different time points | The examination was performed at 1 day, 1 week, 2 weeks, 4 weeks and 8 weeks after intervention.
  A mobility test was performed to evaluate patients' functionality in 2 scenarios: using their best-corrected visual acuity with no LVAs and using the OXSIGHT Smart Glasses. A loop-shaped obstacle course consisting of stationary obstacles from floor to head level was designed for this test.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foster PJ, Johnson GJ. Glaucoma in China: how big is the problem? Br J Ophthalmol. 2001 Nov;85(11):1277-82. doi: 10.1136/bjo.85.11.1277. PMID 11673287
- [Result] Quigley HA, Broman AT. The number of people with glaucoma worldwide in 2010 and 2020. Br J Ophthalmol. 2006 Mar;90(3):262-7. doi: 10.1136/bjo.2005.081224. PMID 16488940
- See also: The Number of People With Glaucoma Worldwide in 2010 and 2020 — https://pubmed.ncbi.nlm.nih.gov/16488940/?from_term=The+number+of+people+with+glaucoma+worldwide+in+2010+and+2020%5B
- See also: Glaucoma in China: How Big Is the Problem? — https://pubmed.ncbi.nlm.nih.gov/11673287/?from_single_result=Johnson+G+J+.+Glaucoma+in+China%3A+how+big+is+the+problem%3F%5BJ%5D.+Br+J+Ophthalmol%2C&expanded_search_query=Johnson+G+J+.+Glaucoma+in+China%3A+how+big+is+the+problem%3F%5BJ%5D.+Br+J+Ophthalmol%2C